CLINICAL TRIAL: NCT00629252
Title: The Effect of Sertindole on Sensory Gating and Cognition in Schizophrenic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough subjects have been recruited in the expected period.
Sponsor: University of Zurich (Other)
Collaborators: University Hospital of Psychiatry, Department Neuropsychopharmacology and Brain Imaging (Other); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 98_PPI-P50; E-11/2007; 2007DR1253
Record Dates: First submitted 2008-01-21; First posted 2008-03-05 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PPI; P50; CANTAB; sensory gating; Schizophrenic patients according to DSM-IV
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Risperidone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Schizophrenic patients treated with sertindole
  Interventions: Drug: Sertindole
- 2 (Active Comparator): Schizophrenic patients treated with risperidone
  Interventions: Drug: Risperidone
- 3 (No Intervention): Healthy controls without any treatment.

INTERVENTIONS:
Drug: Sertindole — oral 12-20 mg/day
  Arms: 1
Drug: Risperidone — oral 2-6mg / day
  Arms: 2

SUMMARY:
This study aims to investigate whether the atypical antipsychotic and mixed 5-HT2/D2 antagonist sertindole modulates or improves both subcortical and cortical information processing in schizophrenic patients who had not or insufficiently responded to previous antipsychotic medication. This goal shall be accomplished by investigating the effect of sertindole of both prepulse inhibition of the acoustic startle (PPI) and P50 suppression of auditory evoked potentials in schizophrenic patients. These effects shall be compared to the effect of risperidone and shall also be compared to untreated healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to DSM IV
* Selected and treated in respect of the SPC (20 mg Serdolect max. and population at risk will be excluded)

Exclusion Criteria:

* DSM IV Axis I disorders other than schizophrenia: Substance-dependence (excepting nicotine-dependence and substance-abuse), recent (2 months) DSM IV diagnosis according to DIA-X of a major affective, anxiety disorder, eating-disorder.
* DSM IV Axis II disorders: Lifetime DSM IV diagnosis of personality disorder.
* ECG: QTc-interval >450 msec.
* Systolic blood pressure <100 mmHg
* Bradycardia (Hf < 50/Min) und Arrhythmias
* Hypokalemia or Hypomagnesemia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
sensory (EEG: P50 suppression) and sensorimotor gating (EMG: PPI) | Before and six weeks after antipsychotic treatment

SECONDARY OUTCOMES:
Cognitive performances | Before and six weeks after antipsychotic treatment
Psychopathology (PANSS rating) | Before and six weeks after antipsychotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Franz X. Vollenweider, Prof. Dr. med., Principal Investigator — University Hospital of Psychiatry, Department Neuropsychopharmacology and Brain Imaging
Locations (1):
- University Hospital of Psychiatry, Department Neuropsychopharmacology and Brain Imaging, Zurich, Canton of Zurich, Switzerland